CLINICAL TRIAL: NCT00027196
Title: Clinical Correlates of Molecular Defects in Familial Cardiomyopathy
Brief Title: Signs and Symptoms Associated With Molecular Defects in Genetically Inherited Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980100; 98-H-0100
Record Dates: First submitted 2001-11-27; First posted 2001-11-28 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-04

CONDITIONS: Congenital Heart Defect
Keywords: Genetics; Cardiac Diseases; Cardiac Hypertrophy; Sudden Death; Arrhythmias
MeSH Terms: conditions — Heart Defects, Congenital; Heart Diseases; Cardiomegaly; Death, Sudden; Arrhythmias, Cardiac

SUMMARY:
Genetically inherited heart diseases (familial cardiopathies) are conditions affecting the heart passed on to family members by abnormalities in genetic information. These conditions are responsible for many heart related deaths and illnesses.

Researchers are interested in learning more about the specific genetic abnormalities causing heart diseases. In addition, they would like to find out how these abnormal genes can contribute to the development of other medical problems.

In order to do this, researchers plan to study patients and family members of patients diagnosed with genetically inherited heart disease. Those people participating in the study will undergo a variety of tests including blood tests, echocardiograms, and magnetic resonance imaging studies (MRI). These tests will be used to help researchers find the genetic problem causing the familial cardiopathy.

Researchers hope that the information gathered from this study can be used to develop better medical care through early diagnosis, management, and treatment plans.

DETAILED DESCRIPTION:
Familial cardiomyopathies (FC) are important cardiovascular causes of morbidity and mortality that demonstrate both allelic and non-allelic genetic heterogeneity. We propose to perform genetic studies to determine novel molecular causes of FC and to describe their clinical correlates. This will permit: (1) pre-symptomatic diagnosis; (2) definition of cardiac phenotype, disease penetrance; (3) natural history; (4) study of abnormal physiology that is a consequence of the molecular defect; (5) elucidation of specific mechanisms of arrythmias and sudden death; and (6) demonstration and characterization of skeletal muscle involvement.

ELIGIBILITY:
INCLUSION AND EXCLUSION CRITERIA

The subjects will consist of family members who may have inherited FC and spouses that may help in the linkage studies. Family members or spouses who do not wish to participate in the research protocol will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9999999
Dates: Start 1998-04; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fananapazir L, Epstein ND. Prevalence of hypertrophic cardiomyopathy and limitations of screening methods. Circulation. 1995 Aug 15;92(4):700-4. doi: 10.1161/01.cir.92.4.700. No abstract available. PMID 7641346
- [Background] Maron BJ, Bonow RO, Cannon RO 3rd, Leon MB, Epstein SE. Hypertrophic cardiomyopathy. Interrelations of clinical manifestations, pathophysiology, and therapy (1). N Engl J Med. 1987 Mar 26;316(13):780-9. doi: 10.1056/NEJM198703263161305. No abstract available. PMID 3547130
- [Background] Wigle ED, Rakowski H, Kimball BP, Williams WG. Hypertrophic cardiomyopathy. Clinical spectrum and treatment. Circulation. 1995 Oct 1;92(7):1680-92. doi: 10.1161/01.cir.92.7.1680. PMID 7671349